CLINICAL TRIAL: NCT05265728
Title: A Single-Arm, Open-Label, Phase 3 Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of Natalizumab (BG00002) Administered to Japanese Participants With Relapsing-Remitting Multiple Sclerosis Via a Subcutaneous Route of Administration
Brief Title: A Study to Evaluate Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of Natalizumab (BG00002) Administered Subcutaneously to Japanese Participants With Relapsing-Remitting Multiple Sclerosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to sponsor decision, not for efficacy or safety reasons.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101MS330
Record Dates: First submitted 2022-02-23; First posted 2022-03-03 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Natalizumab (Experimental): Participants will receive natalizumab 300 mg SC Q4W for 48 weeks.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Administered as specified in the treatment arm
  Other Names: BG00002; Tysabri

SUMMARY:
The primary objective of this study is to evaluate the efficacy of natalizumab 300 milligrams (mg) subcutaneous (SC) every 4 weeks (Q4W) administrations up to 24 weeks in Japanese participants with relapsing-remitting multiple sclerosis (RRMS).

The secondary objectives of the study are to evaluate other clinical and magnetic resonance imaging (MRI) measures of efficacy of natalizumab 300 mg SC Q4W administrations in Japanese participants with RRMS, to evaluate the safety, tolerability, and immunogenicity of natalizumab 300 mg SC Q4W administrations up to 48 weeks in Japanese participants with RRMS, to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of natalizumab 300 mg SC Q4W administrations up to 24 weeks and for an additional 24 weeks in Japanese participants with RRMS.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have had a diagnosis of RRMS, as defined by the revised 2017 McDonald's criteria. All other possible neurologic diagnoses must have been reasonably excluded by means of laboratory and/or imaging studies, in the opinion of the investigator.
* Must have had an EDSS score between 0.0 and 5.5, inclusive.
* Must have had screening MRI or documentation of an MRI within the participant's medical record within 12 months of the screening visit that revealed 3 or more T2 hyperintense lesions consistent with MS.
* Was born in Japan, and biological parents and grandparents were of Japanese origin.

Key Exclusion Criteria:

* Evidence of current severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 14 days prior to Screening, between screening and baseline visit, or at baseline visit, including but not limited to a fever (temperature > 37.5 degrees Celsius [°C]), new and persistent cough, breathlessness, or loss of taste and/or smell.
* Have close contact within 14 days prior to Day 1 with a SARS-CoV-2 positive individual.
* Diagnosis of primary progressive MS or secondary progressive MS.
* An MS exacerbation (relapse) within 30 days prior to enrolment or, in the opinion of the investigator, the participant not having stabilized from a previous relapse prior to enrolment (Day 1).
* The participant is unable to have a brain MRI scan (e.g., a participant with a metal clip to repair a cerebral aneurysm).
* Previous exposure to natalizumab.

Note: Other protocol specified Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (12):
- Japan (12):
  - Juntendo University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - St.Marianna University Hospital, Kawasaki-shi
  - National Center of Neurology and Psychiatry, Kodaira-shi
  - Kansai Medical University Medical Center, Moriguchi-shi
  - Tokyo Metropolitan Hospital Organization Tokyo Metropolitan Ebara Hospital, Ōta-ku
  - The Kitasato Institute Kitasato University Hospital, Sagamihara-shi
  - National Hospital Organization Hokkaido Medical Center, Sapporo
  - Tohoku Medical and Pharmaceutical University Hospital, Sendai
  - Osaka University Hospital, Suita-shi
  - University of Tsukuba Hospital, Tsukuba
  - Tokyo Women's Medical University Yachiyo Medical Center, Yachiyo-shi

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at multiple investigative sites in Japan from 26 April 2022 to 29 June 2023.
Groups:
- Natalizumab: Participants received natalizumab 300 milligrams (mg), subcutaneous (SC), every 4 weeks (Q4W) for 48 weeks.
Period: Overall Study
Arm/Group | Natalizumab
Started | 21
Completed | 13
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Study Terminated by Sponsor | 5
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who had received at least 1 study treatment injection and had at least 1 post baseline efficacy assessment.
Groups:
- Natalizumab: Participants received natalizumab 300 mg, SC, Q4W for 48 weeks.
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Cumulative Number of New Active Lesions up to Week 24 Identified Using Brain Magnetic Resonance Imaging (MRI) Scans
Description: New active lesions were defined as the sum of gadolinium (Gd)-enhancing lesions and non-enhancing new or newly enlarging T2 hyperintense lesions over a period of 24 weeks.
Time Frame: Up to Week 24
Population: FAS included all participants who had received at least 1 study treatment injection and had at least 1 post baseline efficacy assessment. Here, 'overall number of participants analyzed' signifies the number of participants available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Natalizumab
Number analyzed (Participants) | 19
number of lesions | 0.4 (0.60)
Statistical Analysis 1: Comparison: Natalizumab; Test type: Superiority; Least Square Mean (LS mean) = 0.37, 95% CI 2-sided [0.18 to 0.76] — LS mean (95% Confidence Interval [CI]) lesions were obtained from a Poisson distribution model with no explanatory variables

2. Secondary Outcome: Part 2: Cumulative Number of New Active Lesions up to Week 48 Identified Using Brain MRI Scans
Description: New active lesions were defined as the sum of Gd-enhancing lesions and non-enhancing new or newly enlarging T2 hyperintense lesions over a period of 48 weeks.
Time Frame: Up to Week 48
Population: Week 48 analysis set included all participants in the FAS but excluded participants who withdrew from study due to termination of the study by Sponsor. Here, 'overall number of participants analyzed' signifies the number of participants available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Natalizumab
Number analyzed (Participants) | 13
number of lesions | 3.1 (8.47)
Statistical Analysis 1: Comparison: Natalizumab; Test type: Superiority; Least Square Mean = 3.08, 95% CI 2-sided [0.69 to 13.74] — LS mean (95% CI) lesions were obtained from a Poisson distribution model with no explanatory variables

3. Secondary Outcome: Part 1: Proportion of Participants With Any New Active Lesions at Week 24 Identified Using Brain MRI Scans
Description: New active lesions were defined as the sum of gadolinium-enhancing lesions and non-enhancing new or newly enlarging T2 hyperintense lesions.
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 20
proportion of participants | 0.05

4. Secondary Outcome: Part 2: Proportion of Participants With Any New Active Lesions at Week 48 Identified Using Brain MRI Scans
Description: New active lesions were defined as the sum of Gd-enhancing lesions and non-enhancing new or newly enlarging T2 hyperintense lesions.
Time Frame: At Week 48
Population: Week 48 analysis set included all participants in the full analysis set but excluded participants who withdrew from study due to termination of the study by Sponsor. Here, 'overall number of participants analyzed' signifies the number of participants available for outcome measure analysis.
Measure: Number; unit: proportion of participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 13
proportion of participants | 0.15

5. Secondary Outcome: Change From Baseline in Number of Gd-Enhancing Lesions at Week 24 and Week 48
Time Frame: Baseline, Weeks 24 and 48
Population: FAS included all participants who had received at least 1 study treatment injection and had at least 1 post baseline efficacy assessment. Here, 'number analyzed' signifies the number of participants available for analysis at specified time point.
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
number of lesions
  Baseline | 0.5 (1.44)
  Change at Week 24: number analyzed (Participants) | 20
  Change at Week 24 | -0.6 (1.47)
  Change at Week 48: number analyzed (Participants) | 15
  Change at Week 48 | -0.7 (1.72)

6. Secondary Outcome: Number of Non-enhancing New or Newly Enlarging T2 Hyperintense Lesions at Week 24
Time Frame: At Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Natalizumab
Number analyzed (Participants) | 20
number of lesions | 0.3 (1.34)

7. Secondary Outcome: Number of Non-enhancing New or Newly Enlarging T2 Hyperintense Lesions at Week 48
Time Frame: At Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Natalizumab
Number analyzed (Participants) | 13
number of lesions | 2.1 (6.64)

8. Secondary Outcome: Number of New T1 Hypointense Lesions at Week 24
Time Frame: At Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Natalizumab
Number analyzed (Participants) | 20
number of lesions | 0.0 (0.0)

9. Secondary Outcome: Number of New T1 Hypointense Lesions at Week 48
Time Frame: At Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Natalizumab
Number analyzed (Participants) | 13
number of lesions | 0.2 (0.60)

10. Secondary Outcome: Annualized Relapse Rate (ARR) at Week 24, Week 48 and Week 52
Description: ARR is calculated as the total number of relapses that occurred during the treatment period divided by the total number of participant-years. ARR was analyzed using negative binomial regression model.
Time Frame: At Week 24, Week 48 and Week 52
Population: FAS included all participants who had received at least 1 study treatment injection and had at least 1 post baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: relapses per participant-year
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
relapses per participant-year
  Week 24 | 0.508 [0.129 to 2.005]
  Week 48 | 0.462 [0.087 to 2.457]
  Week 52 | 0.456 [0.083 to 2.506]

11. Secondary Outcome: Proportion of Relapse-Free Participants at Week 24 and Week 52
Description: A multiple sclerosis (MS) relapse was defined as the onset of new or recurrent neurological symptoms lasting at least 24 hours, accompanied by new objective abnormalities on a neurological examination, and not explained solely by non-MS processes such as fever, infection, severe stress, or drug toxicity.
Time Frame: At Week 24 and Week 52
Population: as for outcome 10
Measure: Number; unit: proportion of participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
proportion of participants
  Week 24 | 0.8521
  Week 52 | 0.8521

12. Secondary Outcome: Visual Analog Scale (VAS) Score at Week 24 and Week 48
Description: The participant's global impression of his/her well-being was assessed with a VAS. The instrument ranges from 0 to 100 millimeters (mm), where a score of 0 denotes 'poor' and a score of 100 denotes 'excellent'. Higher scores indicates a better health state.
Time Frame: At Week 24 and Week 48
Population: FAS included all participants who had received at least 1 study treatment injection and had at least 1 post baseline efficacy assessment. Here 'number analyzed' signifies the number of participants available for analysis at a specified time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
mm
  Week 24 | 71.0 (22.35)
  Week 48: number analyzed (Participants) | 15
  Week 48 | 61.5 (22.02)

13. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is defined as any AE that has an onset date and time that is on or after the date and time of the first dose of study treatment, or that has worsened after the date and time of the first dose of study treatment through 84 days after the last dose of study treatment.
Time Frame: From first dose of study drug through 84 days after the last dose of study drug (up to Week 60)
Population: Safety analysis set included all participants who had received at least 1 study treatment injection.
Measure: Number; unit: percentage of participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
percentage of participants
  TEAEs | 95.2
  Serious TEAEs | 4.8

14. Secondary Outcome: Percentage of Participants With Positive Anti-John Cunningham Virus (Anti-JCV) Antibodies
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all participants who had received at least 1 study treatment injection.
Measure: Number; unit: percentage of participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
percentage of participants | 57.1

15. Secondary Outcome: Number of Participants With Injection Site Reactions and Injection Reactions
Time Frame: From first dose of study drug through 84 days after the last dose of study drug (up to Week 60)
Population: Safety analysis set included all participants who had received at least 1 study treatment injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
Participants
  Injection Site Reactions | 3 [NA to NA]
  Injection Reactions | 2 [NA to NA]

16. Secondary Outcome: Percentage of Participants With Positive Anti-Natalizumab Antibodies
Time Frame: Baseline up to Week 48
Population: Immunogenicity analysis set included all participants who had received at least 1 study treatment injection and had at least 1 postbaseline assessment for the specific parameter.
Measure: Number; unit: percentage of participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
percentage of participants | 4.8

17. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score at Week 24 and Week 48
Description: The EDSS is a scale based on standardized neurological examination which comprised of optic, brain stem, pyramidal, cerebellar, sensory and cerebral functions, as well as walking ability. It measures the MS disability status on a scale ranging from 0 (normal) to 10 (death due to MS), with higher scores indicating more disability. A negative change from baseline indicates an improvement in the disability.
Time Frame: Baseline, Week 24 and Week 48
Population: Safety analysis set included all participants who had received at least 1 study treatment injection. Here 'number analyzed' signifies the number of participants available for analysis at a specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.83 (1.544)
  Change at Week 24 | 0.02 (0.536)
  Change at Week 48: number analyzed (Participants) | 15
  Change at Week 48 | -0.13 (0.352)

18. Secondary Outcome: Serum Trough Concentration (Ctrough) of Natalizumab
Time Frame: Pre-dose at Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: Pharmacokinetic (PK) analysis set included all participants who had received at least 1 study treatment injection and had at least 1 measurable serum natalizumab concentration. Here 'number analyzed' signifies the number of participants available for analysis at a specified time point.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
milligrams per liter (mg/L)
  Baseline | 0.0 (0.00)
  Week 4 | 10.6 (6.59)
  Week 8 | 15.1 (10.11)
  Week 12: number analyzed (Participants) | 19
  Week 12 | 18.3 (13.22)
  Week 16: number analyzed (Participants) | 20
  Week 16 | 21.1 (16.12)
  Week 20: number analyzed (Participants) | 19
  Week 20 | 20.7 (15.13)
  Week 24: number analyzed (Participants) | 19
  Week 24 | 23.6 (17.77)
  Week 28: number analyzed (Participants) | 19
  Week 28 | 22.2 (14.01)
  Week 32: number analyzed (Participants) | 15
  Week 32 | 20.0 (15.70)
  Week 36: number analyzed (Participants) | 15
  Week 36 | 22.1 (13.95)
  Week 40: number analyzed (Participants) | 15
  Week 40 | 19.5 (15.31)
  Week 44: number analyzed (Participants) | 14
  Week 44 | 22.5 (14.76)
  Week 48: number analyzed (Participants) | 12
  Week 48 | 24.0 (19.00)

19. Secondary Outcome: Serum Concentration of Natalizumab Between Day 6 and Day 8
Description: One blood sample was collected between Day 6 and Day 8.
Time Frame: Between Day 6 and Day 8
Population: PK analysis set included all participants who had received at least 1 study treatment injection and had at least 1 measurable serum natalizumab concentration.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
mg/L | 29.8 (15.07)

20. Secondary Outcome: Trough Alpha-4 (α4) Integrin Saturation
Time Frame: Pre-dose at Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: Pharmacodynamic (PD) analysis set included all participants who had received at least 1 study treatment injection and had at least 1 assessment for α4-integrin saturation, serum soluble vascular cell adhesion molecule-1 (VCAM-1) concentration, and lymphocyte counts with lymphocyte subsets. Here 'number analyzed' signifies the number of participants available for analysis at a specified time point.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
percentage
  Baseline: number analyzed (Participants) | 20
  Baseline | 4.9 (4.99)
  Week 4 | 81.9 (18.31)
  Week 8 | 82.6 (20.85)
  Week 12: number analyzed (Participants) | 19
  Week 12 | 82.8 (20.22)
  Week 16: number analyzed (Participants) | 20
  Week 16 | 87.3 (19.52)
  Week 20: number analyzed (Participants) | 19
  Week 20 | 87.0 (17.10)
  Week 24: number analyzed (Participants) | 18
  Week 24 | 87.1 (23.59)
  Week 28: number analyzed (Participants) | 19
  Week 28 | 86.4 (21.97)
  Week 32: number analyzed (Participants) | 15
  Week 32 | 87.1 (26.46)
  Week 36: number analyzed (Participants) | 15
  Week 36 | 82.6 (23.93)
  Week 40: number analyzed (Participants) | 15
  Week 40 | 84.6 (26.27)
  Week 44: number analyzed (Participants) | 14
  Week 44 | 83.3 (25.22)
  Week 48: number analyzed (Participants) | 12
  Week 48 | 80.1 (24.98)

21. Secondary Outcome: Serum Soluble VCAM-1 Concentrations
Time Frame: Pre-dose at Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: PD analysis set included all participants who had received at least 1 study treatment of study treatment and had at least 1 assessment for α4-integrin saturation, serum soluble VCAM-1 concentration, and lymphocyte counts with lymphocyte subsets. Here 'number analyzed' signifies the number of participants available for analysis at a specified time point.
Measure: Mean (Standard Deviation); unit: micrograms per liter (µg/L)
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
micrograms per liter (µg/L)
  Baseline | 468.9 (80.90)
  Week 4 | 237.8 (66.29)
  Week 8 | 248.2 (86.47)
  Week 12: number analyzed (Participants) | 19
  Week 12 | 239.8 (77.96)
  Week 16: number analyzed (Participants) | 20
  Week 16 | 231.8 (70.76)
  Week 20: number analyzed (Participants) | 19
  Week 20 | 236.0 (71.22)
  Week 24: number analyzed (Participants) | 19
  Week 24 | 237.4 (80.38)
  Week 28: number analyzed (Participants) | 19
  Week 28 | 229.1 (80.47)
  Week 32: number analyzed (Participants) | 15
  Week 32 | 238.1 (86.11)
  Week 36: number analyzed (Participants) | 15
  Week 36 | 243.1 (105.46)
  Week 40: number analyzed (Participants) | 15
  Week 40 | 235.6 (80.59)
  Week 44: number analyzed (Participants) | 14
  Week 44 | 242.0 (72.06)
  Week 48: number analyzed (Participants) | 12
  Week 48 | 244.1 (87.07)

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 76 weeks; Adverse Events were assessed up to Week 60
Description: Safety analysis set included all participants who had received at least 1 study treatment injection.
Groups:
- Natalizumab: Participants received natalizumab 300 mg SC Q4W for 48 weeks.
Arm/Group | Natalizumab
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=21)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=21)
Dental caries (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Injection site reaction (General disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 2
Covid-19 (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Lymphocyte count increased (Investigations) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Menstrual headache (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally, the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor's Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of the Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT05265728/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT05265728/SAP_001.pdf